CLINICAL TRIAL: NCT03062293
Title: Newcastle Low Back Pain Intervention Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Northumbria University (Other)
Collaborators: European Space Agency (Other); The University of Queensland (Other); International Space University (Unknown); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRED2016
Record Dates: First submitted 2016-10-11; First posted 2017-02-23 (Actual); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Low Back Pain, Mechanical
Keywords: Lumbo-pelvic muscles; Rehabilitation; Exercise; Low back pain; Functional Re-adaptive Exercise Device
MeSH Terms: conditions — Low Back Pain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Repeat measures within subject design
Masking Description: Ultrasound image time points are blinded to the assessor by a party not involved in the study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Functional Re-adaptive Exercise Device (Experimental): Single arm for within subject repeated measures design.
  Interventions: Device: Functional Re-adaptive Exercise Device

INTERVENTIONS:
Device: Functional Re-adaptive Exercise Device — Exercise intervention 3 times per week for up to 30min. Difficulty and time will be progressed as indicated by clinical presentation, assessed by the Physiotherapist team.
  Other Names: FRED

SUMMARY:
The aim of this study is to investigate if six-weeks of exercise intervention, 3 times per week on the Functional Re-adaptive Exercise Device (FRED) reduces non-specific mechanical low back pain in adults ages 18-60.

DETAILED DESCRIPTION:
The aim of this study is to investigate whether an six-week FRED exercise intervention reduces low back pain (LBP) and improves a range of related outcomes.

The objectives of this study are to examine

1. whether FRED exercise reduces mechanical LBP ( low back pain);
2. whether FRED exercise improves functional and static balance in people with LBP;
3. whether FRED exercise has an effect on cross-sectional area (CSA) of relevant lumbo-pelvic muscles;
4. whether FRED exercise has an effect on TrA (Transversus Abdominis), LM ( Lumbar Multifidus), lumbar Erector Spinae, External and Internal Oblique muscle activity and function in individuals with LBP;
5. whether FRED exercise has an effect on TrA and internal oblique muscle thickness;
6. the rate of muscle physiology change in response to FRED exercise in people with LBP;
7. whether FRED exercise affects the analgesic intake, need for intervention and physical activity level of individuals with LBP;
8. whether FRED exercise affects wellbeing and every-day function in people with LBP;
9. the rate of change of level of pain, wellbeing and of function (incl. balance) in response to FRED exercise in people with LBP.

ELIGIBILITY:
Inclusion Criteria:

* Mechanical LBP for 8 weeks or longer
* Score of < 15 on FABQ
* Age 18-60
* Commitment to taking part in the study for its full duration

Exclusion Criteria:

* Presence of "red flags" - indicative of non-mechanical LBP
* Score of > 15 on FABQ or other indicators of a likely poor response to a solely physical approach to treatment incl. seeking compensation for LBP
* Exercise contraindicated as per Physical Activity Readiness Questionnaire
* Inability to exercise safely on the FRED
* Pregnancy
* Surgery within the previous nine months
* Difficulty to exercise safely in standing for 30 mins 3x/week
* Cardio/respiratory disease
* Neurological disorders
* BMI > 28 where adipose tissue infringes on ultrasound imaging and intramuscular electrode placement

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Change in Intramuscular EMG of Lumbo-pelvic muscles | within 1 week prior to intervention, and within 1 week post intervention (2 data collection
  iEMG of Lumbar Multifudus (LM), Transversus Abdominus (TrA), External Obliques and Internal obliques during exercise and balance tasks

SECONDARY OUTCOMES:
Change in muscular arcitecture via Ultrasound imaging | At baseline (intervention -6 weeks) within 1 week prior to intervention, within 1 week post intervention, 1 x week during intervention, and at intervention +12 weeks (10 data collections)
  USI of cross sectional area and thickness of Lumbar Multifudus (LM),and thickness of Transversus Abdominus (TrA)
VICON/ force plate kinematic data | within 1 week prior to intervention and and within 1 week post intervention (2 data collections)
  Measuring postural sway changes in center of pressure during the balance and rapid arm movement tasks, repeated measure throughout study
Participant Activity Log | Daily from baseline data collection to intervention +16 weeks follow-up (total 203 days)
SF-36 II . | At baseline (intervention -6 weeks) within 1 week prior to intervention, within 1 week post intervention, at intervention +6 week, +12 weeks and +16 weeks follow up (5 data collections)
  Version 2, UK, acute recall
Patient Specific Functional Scale | At baseline (intervention -6 weeks) within 1 week prior to intervention, within 1 week post intervention, at intervention +6 week, +12 weeks and +16 weeks follow up (5 data collections)
  repeated measure throughout study
Numeric Rating Scale for Pain | At baseline (intervention -6 weeks) within 1 week prior to intervention, within 1 week post intervention, at intervention +6 week, +12 weeks and +16 weeks follow up (5 data collections)

OTHER OUTCOMES:
Movement variability during exercise | At baseline (intervention -6 weeks) within 1 week prior to intervention, within 1 week post intervention, 3 x week during intervention, at intervention +6 weeks and +12 weeks follow up (22 data collections)
  Changes in neuromuscular control during FRED exercise

IPD SHARING:
Plan to Share IPD: No
NO IPD will be available to researchers outside of the research team.

REFERENCES:
- [Background] Caplan, N, Gibbon, KC, Hibbs, A & Debuse, D 2014, 'Phasic-to-tonic shift in tunk muscle activity during low-impact weight bearing exercise', Acta Astronautica, vol 104, pp. 388-395.
- [Background] Debuse D, Birch O, St Clair Gibson A, Caplan N. Low impact weight-bearing exercise in an upright posture increases the activation of two key local muscles of the lumbo-pelvic region. Physiother Theory Pract. 2013 Jan;29(1):51-60. doi: 10.3109/09593985.2012.698718. Epub 2012 Jul 12. PMID 22789062
- [Background] Gibbon KC, Debuse D, Caplan N. Low impact weight-bearing exercise in an upright posture achieves greater lumbopelvic stability than overground walking. J Bodyw Mov Ther. 2013 Oct;17(4):462-8. doi: 10.1016/j.jbmt.2013.02.004. Epub 2013 Apr 22. PMID 24139004
- [Background] Evetts SN, Caplan N, Debuse D, Lambrecht G, Damann V, Petersen N, Hides J. Post space mission lumbo-pelvic neuromuscular reconditioning: a European perspective. Aviat Space Environ Med. 2014 Jul;85(7):764-5. doi: 10.3357/asem.3943.2014. PMID 25022167